CLINICAL TRIAL: NCT00421551
Title: A Randomized Multicenter Study With Non-inferiority Hypothesis, Comparing the Availability to Maintain a Complete Viral Suppression by a Monotherapy of Darunavir/r to a NRTI Containing Regimen Including Darunavir/r, in HIV-1 Infected Patients With Previous Prolonged Complete Viral Suppression. ANRS 136 MONOI
Brief Title: Study Comparing Efficacy and Safety of Darunavir Boosted With Ritonavir to HART With 2 NRTI and Darunavir Boosted With Ritonavir in HIV-1 Infected Patients ANRS136
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Collaborators: Tibotec Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Organization: ANRS, Emerging Infectious Diseases (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006-005962-38; ANRS 136 MONOI
Record Dates: First submitted 2007-01-11; First posted 2007-01-12 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2013-07

CONDITIONS: HIV Infections
Keywords: HIV Infections; darunavir; Ritonavir; HIV Protease Inhibitors; treatment experienced
MeSH Terms: conditions — HIV Infections | interventions — Darunavir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Darunavir; Drug: ritonavir
- 2 (Active Comparator)
  Interventions: Drug: Darunavir; Drug: ritonavir

INTERVENTIONS:
Drug: Darunavir — during the 48 first weeks of the trial, (2x300mg) twice a day between W48 and W96, (2x400mg) once a day
  Other Names: Prezista
Drug: ritonavir — during the first 48 weeks, 100mg twice a day between W48 and W96, 100mg once a day
  Other Names: Norvir

SUMMARY:
The purpose of this study is to evaluate whether a monotherapy of boosted darunavir is able to maintain the virological success until 48 weeks in comparison to a standard therapy 2 INTI + darunavir/r in HIV infected patients with full viral suppression.

DETAILED DESCRIPTION:
The chronicity of the disease which will require treatment over decades, long-term adverse events associated with standard combined antiretroviral therapy, emphasize the need for simpler, alternative treatment strategies for HIV infection. The goal of antiretroviral therapy in 2006 is the durability of treatment with less toxicity and reduced exposure to drugs. Previous studies have shown that single boosted PI maintenance therapy such as lopinavir (LPV/r), were effective in maintaining virological efficacy. Furthermore, in case of virological failure, limited resistance has been described. darunavir/r, a new PI, has been shown to be highly potent, exhibits a high genetic barrier to resistance and appears to be well tolerated. This study aimed to evaluate whether darunavir/r can represent a potential strategy therapeutic as single therapy in patients who have full virologic suppression At entry, subjects with HIV RNA below 50 cp/ml switch from their current therapy which can be 2 NRTI and IP, 2 NRTI and NNRTI, 3 NRTI to darunavir/r with their 2 NRTIs for 8 weeks (Phase I). If patients remain below 50 cp/ml and has no intolerance to darunavir at week -4, they are included in the phase II and will be randomized either to receive darunavir/r alone or to continue 2 NRTI and darunavir/r for until W48 (Phase II). Patients will be monitored at W4, W8 and then every 8 weeks until W48 for the primary endpoint. To evaluate the durability and safety of this strategy, patients will be followed up to W96

ELIGIBILITY:
Inclusion Criteria:

* Confirmed HIV-1 infection.
* Documented level of HIV-1 RNA at initiation of antiretroviral treatments
* Prior antiretroviral regimen, including at least 2 NRTIs combined to 1 PI or NNRTI or a third NRTI for at least 18 months prior to study entry.
* CD4 count of 200 cells per mm3 or greater.
* Viral load below 400 copies per ml within 18 months prior to entry and below 50 copies per mL at entry.
* Willing to use acceptable methods of contraception

Exclusion Criteria:

* Previous virological failure under prior PI-based regimen.
* Prior therapy in the darunavir.
* HIV-2 infected patients.
* Absence of documented level of HIV-1 RNA at initiation of antiretroviral treatments
* Hepatitis B or C infection within 90 days prior to study entry.
* Therapies including interferon, interleukin-2, cytotoxic chemotherapy or immunosuppressors at study entry.
* Serious acute illness requiring systemic treatment or hospitalization in the 14 days prior to study entry.
* Treatment for an active AIDS defining opportunistic infection within 30 days prior to screening
* Drug or alcohol use or any dependence that would interfere with compliance.
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2007-03; Primary Completion 2010-06 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with virological success, the virological failure is defined as 2 consecutive plasma viral load measurements greater or equal to 400 cp/ml within 2 weeks at W48 | W48

SECONDARY OUTCOMES:
Proportion of patients with virological success between W48 and W96, | W96
Proportion of patients with HIV-1 RNA below 50 copies/mL, between 50 to 400 copies/mL and > 400 copies/ml from D0 to W96, | W96
Time to virologic failure, | between W0 and W96
PI genotypic resistance mutations occurring during the follow-up | between W0 and W96
Change in proviral DNA at D0, W48 and W96, | W0, W48 and W96
Change in CD4 count from D0 to W96. | D0, W96
Comparing plasma HIV-1 RNA genotypic resistance with DNA genotypic resistance at entry | D0
Quantification of HIV RNA in the genital compartment between D0 and W48 (sub-study with 40 patients enrolled, 20 patients in each arm of strategy). | D0 and W48
Incidence of clinical endpoints | W96
Modification of treatment strategies and withdrawal of study treatment. | between D0 and W96
Tolerance of Darunavir (Grade 3 and 4 laboratory abnormalities and signs and symptoms). | between D0 and W96
Change in lipidic and glucidic profile and distribution of fat tissue by DEXA-scan (sub-study in 160 patients enrolled). | W0, W48 and W96
Self-reported adherence and symptom self-evaluation. | W0, W4, W24, W48, W96
The proportion of patients with HIV RNA below 50 copies/mL in darunavir/r monotherapy arm after resuming 2 previous NRTIs in case of virological failure. | between W0 and W96
Search for predictive factors of virological failure (level of proviral DNA, Cmin LPV, …). | between W0 and W96
evaluation of the mineral bone density by DEXA-scan (sub-study in 160 patients enrolled). | W96

CONTACTS AND LOCATIONS:
Overall Officials: Christine Katlama, MD, Principal Investigator — AP-HP hopital Pitié salpetriere Paris; Philippe Flandre, Study Chair — Inserm UMR S720
Locations (1):
- Service des maladies infectieuses et tropicales Hopital Pitie salpetriere, Paris, France

REFERENCES:
- [Derived] Lambert-Niclot S, Grude M, Meynard JL, Marcelin AG, Valantin MA, Flandre P, Izopet J, Moinot L, Bouteloup V, Calvez V, Katlama C, Girard PM, Morand-Joubert L. Ultrasensitive Human Immunodeficiency Virus Type 1 Viral Load as a Marker of Treatment Choice for Simplification Strategies. Clin Infect Dis. 2018 Nov 28;67(12):1883-1889. doi: 10.1093/cid/ciy382. PMID 29767684
- [Derived] Lambert-Niclot S, Flandre P, Valantin MA, Soulie C, Fourati S, Wirden M, Sayon S, Pakianather S, Bocket L, Masquelier B, Dos Santos G, Katlama C, Calvez V, Marcelin AG. Similar evolution of cellular HIV-1 DNA level in darunavir/ritonavir monotherapy versus triple therapy in MONOI-ANRS136 trial over 96 weeks. PLoS One. 2012;7(7):e41390. doi: 10.1371/journal.pone.0041390. Epub 2012 Jul 25. PMID 22848481
- [Derived] Katlama C, Valantin MA, Algarte-Genin M, Duvivier C, Lambert-Niclot S, Girard PM, Molina JM, Hoen B, Pakianather S, Peytavin G, Marcelin AG, Flandre P. Efficacy of darunavir/ritonavir maintenance monotherapy in patients with HIV-1 viral suppression: a randomized open-label, noninferiority trial, MONOI-ANRS 136. AIDS. 2010 Sep 24;24(15):2365-74. doi: 10.1097/QAD.0b013e32833dec20. PMID 20802297